CLINICAL TRIAL: NCT06517134
Title: Association Between GP Characteristics and Prescription Patterns for Antihypertensive Drugs: A Cross-sectional Study in Normandy, France
Brief Title: Prescribing Patterns of Antihypertensive Drugs in Uncomplicated Hypertension
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Xavier HUMBERT, Assistant professor of general practice, University Hospital, Caen
Other Study IDs: 24-01
Record Dates: First submitted 2024-07-19; First posted 2024-07-24 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Hypertension,Essential; Cardiovascular Diseases
Keywords: hypertension; prescriptions; primary care
MeSH Terms: conditions — Essential Hypertension; Cardiovascular Diseases; Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypertensive subjects
  Interventions: Drug: Antihypertensive Agents
- non-hypertensive subjects

INTERVENTIONS:
Drug: Antihypertensive Agents — use of antihypertensive drugs
  Groups: hypertensive subjects

SUMMARY:
Hypertension incurs substantial cardiovascular morbidity and mortality, particularly in primary prevention settings. General practitioners (GPs) play a pivotal role in the management of hypertension in primary care, yet variations exist among GPs. The determinants shaping GPs' antihypertensive medication (AD) prescription patterns in the setting of hypertension remain ambiguous. This investigation sought to elucidate how GPs' characteristics and professional activities influence AD prescriptions. A cross-sectional study utilizing a sample of 2,165 GPs was conducted in Normandy, France, in 2019. The ratio of AD prescriptions to overall prescription volume was computed for each practitioner. GPs were classified as 'low' or 'high' AD prescribers based on the median of this ratio. The ratio was examined in relation to GPs' demographic and professional variables such as age, gender, practice setting, years of experience, consultation frequency, the demographics and socioeconomic status of their patient panels, and prevalence of chronic conditions in patients. These associations were explored using both univariate and multivariate analyses.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had at least one visit to their GP in 2019 were included, but minors were omitted.

Exclusion Criteria:

* minors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participant pool for this study comprised GP characteristics and prescription practices within the Normandy region in northwestern France during the course of 2019. With a resident population of 3,325,032 as of January 1, 2019, and a total of 2,165 registered GPs, the study was well-situated to offer a representative analysis.
  In order to focus on conventional full-time primary GP care, practitioners whose primary professional focus included specialties such as osteopathy, acupuncture, homeopathy, or nutrition were excluded. Furthermore, GPs with fewer than 300 annual consultations/visits (less than one per day), fewer than 2,000 annual drug prescriptions, no patients with any of the 30 chronic diseases that qualify for no-charge treatment under French law, or solely very low-income patients (eligible for no-charge GP visits as defined by French legislation) were also excluded.
Sampling Method: Non-Probability Sample
Enrollment: 3325032 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
GP demographics | 1 year
  age and gender of GPs, the urban or rural classification of the practice location (based on the GP's clinic postal code and DATASANTE tables from the French National Institute for Statistics and Economic Studies, INSEE), and the number of years in practice.
medical practice activities | 1 year
  frequency of home visits and consultations, the total number of registered patients, the average number of visits or consultations per patient, the average patient age, the number of very low-income patients, and the prevalence of registered chronic diseases (notably diabetes mellitus and cardiovascular diseases).

CONTACTS AND LOCATIONS:
Locations (1):
- Xavier Humbert, Caen, France

IPD SHARING:
Plan to Share IPD: No